CLINICAL TRIAL: NCT03538821
Title: The Effects of a Daily Intake of Protein From Cod Fillet and Cod Residual Material for 8 Weeks on Serum Lipids and Fatty Acids, Glucose Regulation and Inflammation Markers in Overweight or Obese Adults: A Randomized Controlled Trial.
Brief Title: The Effects of Intake of Protein From Cod Fillet and Cod Residual Material on Lipid Regulation, Glucose Regulation and Inflammation in Overweight or Obese Adults.
Acronym: COD2017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other); K. Halstensen AS (Unknown); Regional Research Fund Western Norway (Unknown); Nofima (Other)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, Researcher, PhD, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015/75 part 1
Record Dates: First submitted 2018-05-14; First posted 2018-05-29 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Overweight and Obesity; Healthy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intact cod protein from fillet (Experimental): Dietary supplement: intact cod protein from fillet, 8 g protein daily for 8 weeks
  Interventions: Dietary Supplement: Intact cod protein from fillet
- Intact cod protein from residual material (Experimental): Dietary supplement: intact cod protein from residual material, 8 g protein daily for 8 weeks
  Interventions: Dietary Supplement: Intact cod protein from residual material
- Control (Experimental): Control group receive tablet containing fillers and no proteins
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Intact cod protein from fillet — Intact cod protein from fillet 8 g protein daily for 8 weeks
  Arms: Intact cod protein from fillet
Dietary Supplement: Intact cod protein from residual material — Intact cod protein from residual material, 8 g protein daily for 8 weeks
  Arms: Intact cod protein from residual material
Dietary Supplement: Control — Control group receive tablet containing fillers
  Arms: Control

SUMMARY:
A high intake of fish is associated with positive health effects, including prevention and treatment of chronic non-communicable diseases, such as cardiovascular diseases (CVDs) and type 2 diabetes. These health effects have traditionally been attributed to the omega-3 fatty acids in fatty fish, but recent studies have suggested that also fish proteins may improve biomarkers of metabolic disease. Intake of cod fillet have previously shown beneficial effects on blood lipids, glucose regulation and body composition in adults with overweight or obesity. Health effect of cod residual material from fillet production (i.e., head, backbone, skin, cutoffs and entrails) have so far not been investigated, but residuals from other fish species have shown promising effects on glucose regulation in rats. The main aim of the current study is to investigate the effects of protein from cod fillet and cod residuals on serum lipids, glucose regulation and inflammatory markers in healthy overweight or obese adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27 kg/m2
* Fasting blood glucose ≤7 mmol/L
* Physically inactive
* Percent body fat > 25 % for men and > 35 % for women

Exclusion Criteria:

* Allergies towards fish, milk, egg, gluten
* Tobacco use > 10 cigarettes (or snus) per day
* Diseases affecting the heart, intestinal function, kidney function or insulin secretion
* Medications targeting cholesterol -or glucose metabolism, hypertension
* Use of dietary supplements
* Pregnancy or lactation

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Biomarkers related to lipid metabolism | 8 weeks
  Lipids will be measured in fasting serum samples

SECONDARY OUTCOMES:
Biomarkers related to glucose regulation | 8 weeks
  Glucose, insulin and GLP-1 and will be measured in serum/plasma sampled in fasting and postprandial conditions.
Inflammatory markers | 8 weeks
  Cytokines will be measured in fasting serum/plasma
Body composition | 8 weeks
  Percent body fat will be measured using bioimpedance

CONTACTS AND LOCATIONS:
Locations (1):
- Oddrun Anita Gudbrandsen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vikoren LA, Nygard OK, Lied E, Rostrup E, Gudbrandsen OA. A randomised study on the effects of fish protein supplement on glucose tolerance, lipids and body composition in overweight adults. Br J Nutr. 2013 Feb 28;109(4):648-57. doi: 10.1017/S0007114512001717. Epub 2012 May 31. PMID 22647247
- [Background] Drotningsvik A, Mjos SA, Pampanin DM, Slizyte R, Carvajal A, Remman T, Hogoy I, Gudbrandsen OA. Dietary fish protein hydrolysates containing bioactive motifs affect serum and adipose tissue fatty acid compositions, serum lipids, postprandial glucose regulation and growth in obese Zucker fa/fa rats. Br J Nutr. 2016 Oct;116(8):1336-1345. doi: 10.1017/S0007114516003548. Epub 2016 Oct 18. PMID 27751188